CLINICAL TRIAL: NCT00977080
Title: The IMPACT SHPT Study: Study to Evaluate the Improved Management of iPTH With Paricalcitol-centered Therapy vs. Cinacalcet Therapy With Low-dose Vitamin D in Hemodialysis Patients With Secondary Hyperparathyroidism
Brief Title: Evaluation of the Effectiveness of Paricalcitol Versus Cinacalcet With Low-Dose Vitamin D
Acronym: IMPACT SHPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-967; 2009-011378-14 (EudraCT Number)
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism; Hemodialysis
Keywords: Zemplar; paricalcitol; IMPACT SHPT; Hemodialysis; Chronic Kidney Disease Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — paricalcitol; Cinacalcet; 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IV Paricalcitol (Active Comparator): Participants in the IV stratum received intravenous (IV) paricalcitol and, if hypercalcemia (calcium >= 10.5 mg/dL), received 30 mg of oral cinacalcet. Paricalcitol was dosed at 0.07 mcg/kg with titration every 2 weeks.
  Interventions: Drug: Paricalcitol
- Cinacalcet (at sites with IV paricalcitol) (Active Comparator): Participants in the IV stratum received 30 mg of oral cinacalcet daily with a low-dose vitamin D receptor activator (VDRA) (doxercalciferol IV 1 mcg 3 times weekly (TIW) at sites in the US and alfacalcidol capsules 0.25 mcg daily at sites in Russia).
  Interventions: Drug: Cinacalcet
- Oral paricalcitol (Active Comparator): Participants in the oral stratum received oral paricalcitol and, if hypercalcemia (calcium >= 10.5 mg/dL), received 30 mg of oral cinacalcet. Paricalcitol was dosed at mcg = IPTH/60 3 times weekly (TIW) with titration every 2 weeks.
  Interventions: Drug: Paricalcitol
- Cinacalcet (at sites with oral paricalcitol) (Active Comparator): Participants in the oral stratum received 30 mg of oral cinacalcet daily with a low-dose vitamin D receptor activator (VDRA) (alfacalcidol capsules 0.25 mcg daily).
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol dosed per label by region (participants were to receive cinacalcet if they developed hypercalcemia)
  Other Names: ABT-358; Zemplar
  Arms: IV Paricalcitol; Oral paricalcitol
Drug: Cinacalcet — On-label oral cinacalcet by region with low dose vitamin D receptor activator (VDRA) (either doxercalciferol at US sites or alfacalcidol at non-US sites)
  Other Names: Sensipar; Mimpara; Hectorol
  Arms: Cinacalcet (at sites with IV paricalcitol); Cinacalcet (at sites with oral paricalcitol)

SUMMARY:
Evaluates the effectiveness of on-label Paricalcitol versus Cinacalcet with Low-Dose Vitamin D.

DETAILED DESCRIPTION:
During a 4-week washout period, participants stopped taking cinacalcet or other vitamin D receptor activators (VDRAs). (Participants who were naive to cinacalcet or VDRAs did not have to wash out). At randomization, participants entered a 28-week open-label treatment period, during which they received either cinacalcet or paricalcitol. Participants who were assigned to receive paricalcitol were dosed according to the approved label in their respective geographic regions (i.e., IV at sites in the US and Russia and oral at sites in Europe). Supplemental cinacalcet was administered to participants in the paricalcitol arms who developed hypercalcemia (defined as >= 10.5 mg/dL). The evaluation period was from Weeks 21 to 28.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients >= 18 years old.
2. Patient was diagnosed with Stage 5 chronic kidney disease (CKD) and had been receiving intravenous (IV) or oral vitamin D receptor activators (VDRAs) or cinacalcet during the 8 weeks prior to the screening period or naïve patients who had not received VDRA or cinacalcet within 8 weeks of screening.
3. Patient was on maintenance HD (hemodialysis) 3 times weekly (TIW) for at least 3 months prior to screening and was expected to remain on HD for the duration of the study.
4. For entry into the Pre-Treatment Washout Period (for patients who were not naïve to VDRAs and cinacalcet), the patient had to have screening laboratory values of:

   * iPTH level 130 to 700 pg/mL
   * Serum Total Alkaline Phosphatase level >= 40 U/L
   * Calcium level <= 10.0 mg/dL (2.49 mmol/L)
   * Calcium-phosphorus product (CaxP) <= 75 mg2/dL2 (US) and <= 70 mg2/dL2 (non-US)

Exclusion Criteria

1. Patient had a history of parathyroidectomy.
2. Patient had a current malignancy (with the exception of basal or squamous cell carcinoma of the skin), or clinically significant liver disease, in the opinion of the investigator.
3. Use of known inhibitors (i.e., ketoconazole) or inducers (i.e., carbamazepine) of cytochrome P450 (including grapefruit and/or grapefruit juice) 3A (CYP3A) or drugs metabolized by cytochrome P450 2D6 (CYP2D6) (e.g., flecainide, vinblastine, thioridazine, and most tricyclic antidepressants) within 2 weeks prior to study drug administration. Commonly used beta blockers such as metoprolol and carvedilol are allowed but are metabolized by CYP2D6; thus, an adjustment to a lower dose may have been required.
4. Patient was known to be human immunodeficiency (HIV) positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samina Khan, MD, Study Director — Abbott
Locations (83):
- United States (30):
  - Site Reference ID/Investigator# 22781, Tempe, Arizona
  - Site Reference ID/Investigator# 24342, Chula Vista, California
  - Site Reference ID/Investigator# 21142, Los Angeles, California
  - Site Reference ID/Investigator# 22762, Los Angeles, California
  - Site Reference ID/Investigator# 22758, Riverside, California
  - Site Reference ID/Investigator# 21442, San Diego, California
  - Site Reference ID/Investigator# 23688, Arvada, Colorado
  - Site Reference ID/Investigator# 21370, Coral Springs, Florida
  - Site Reference ID/Investigator# 25902, Hudson, Florida
  - Site Reference ID/Investigator# 21146, Lauderdale Lakes, Florida
  - Site Reference ID/Investigator# 26743, Lauderdale Lakes, Florida
  - Site Reference ID/Investigator# 22788, Miami, Florida
  - Site Reference ID/Investigator# 22722, Orlando, Florida
  - Site Reference ID/Investigator# 23147, Tampa, Florida
  - Site Reference ID/Investigator# 22778, Meridian, Idaho
  - Site Reference ID/Investigator# 21369, Detroit, Michigan
  - Site Reference ID/Investigator# 22786, Detroit, Michigan
  - Site Reference ID/Investigator# 21144, St Louis, Missouri
  - Site Reference ID/Investigator# 21443, St Louis, Missouri
  - Site Reference ID/Investigator# 21145, Omaha, Nebraska
  - Site Reference ID/Investigator# 22505, Flushing, New York
  - Site Reference ID/Investigator# 22759, Toledo, Ohio
  - Site Reference ID/Investigator# 22796, Lancaster, Pennsylvania
  - Site Reference ID/Investigator# 22770, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 22772, Aiken, South Carolina
  - Site Reference ID/Investigator# 21147, Orangeburg, South Carolina
  - Site Reference ID/Investigator# 22982, Houston, Texas
  - Site Reference ID/Investigator# 21143, Houston, Texas
  - Site Reference ID/Investigator# 22506, San Antonio, Texas
  - Site Reference ID/Investigator# 22776, Bluefield, West Virginia
- Czechia (3):
  - Site Reference ID/Investigator# 22311, Brno
  - Site Reference ID/Investigator# 22310, Jilemnice
  - Site Reference ID/Investigator# 21624, Ústí nad Labem
- Denmark (4):
  - Site Reference ID/Investigator# 22363, Aalborg
  - Site Reference ID/Investigator# 23105, Copenhagen
  - Site Reference ID/Investigator# 23909, Fredericia
  - Site Reference ID/Investigator# 22462, Holstebro
- Germany (6):
  - Site Reference ID/Investigator# 21748, Coburg
  - Site Reference ID/Investigator# 33268, Darmstadt
  - Site Reference ID/Investigator# 35903, Düsseldorf
  - Site Reference ID/Investigator# 21742, Frankfurt
  - Site Reference ID/Investigator# 21744, Heilbronn
  - Site Reference ID/Investigator# 21368, Lüdenscheid
- Greece (6):
  - Site Reference ID/Investigator# 22362, Athens
  - Site Reference ID/Investigator# 38970, Thessaloniki
  - Site Reference ID/Investigator# 22322, Thessaloniki
  - Site Reference ID/Investigator# 22463, Thessaloniki
  - Site Reference ID/Investigator# 22323, Thessaloniki
  - Site Reference ID/Investigator# 39262, Thessaloniki
- Italy (6):
  - Site Reference ID/Investigator# 22312, Bergamo
  - Site Reference ID/Investigator# 21746, Genova
  - Site Reference ID/Investigator# 39180, Lucca
  - Site Reference ID/Investigator# 22314, Milan
  - Site Reference ID/Investigator# 21367, Pavia
  - Site Reference ID/Investigator# 21745, Pesaro
- Netherlands (3):
  - Site Reference ID/Investigator# 21842, Alkmaar
  - Site Reference ID/Investigator# 22309, Delft
  - Site Reference ID/Investigator# 21843, Dordrecht
- Portugal (4):
  - Site Reference ID/Investigator# 38903, Beja
  - Site Reference ID/Investigator# 38531, Faro
  - Site Reference ID/Investigator# 22464, Lisbon
  - Site Reference ID/Investigator# 23910, Vila Franca de Xira
- Russia (2):
  - Site Reference ID/Investigator# 24643, Moscow
  - Site Reference ID/Investigator# 24642, Moscow
- Spain (9):
  - Site Reference ID/Investigator# 21361, Barcelona
  - Site Reference ID/Investigator# 21364, Córdoba
  - Site Reference ID/Investigator# 22366, L'Hospitalet, Barcelona
  - Site Reference ID/Investigator# 38343, Madrid
  - Site Reference ID/Investigator# 21362, Madrid
  - Site Reference ID/Investigator# 21363, Palma de Mallorca
  - Site Reference ID/Investigator# 22367, Pamplona
  - Site Reference ID/Investigator# 38462, Puerto de la Cruz
  - Site Reference ID/Investigator# 21365, Seville
- Sweden (3):
  - Site Reference ID/Investigator# 23913, Linköping
  - Site Reference ID/Investigator# 23782, Stockholm
  - Site Reference ID/Investigator# 22364, Uppsala
- United Kingdom (7):
  - Site Reference ID/Investigator# 23912, Birmingham
  - Site Reference ID/Investigator# 21747, Coventry
  - Site Reference ID/Investigator# 23102, London
  - Site Reference ID/Investigator# 23104, London
  - Site Reference ID/Investigator# 23103, Manchester
  - Site Reference ID/Investigator# 41982, Omagh, Northern Ireland
  - Site Reference ID/Investigator# 40222, Sheffield

REFERENCES:
- [Derived] Cozzolino M, Ketteler M, Martin KJ, Sharma A, Goldsmith D, Khan S. Paricalcitol- or cinacalcet-centred therapy affects markers of bone mineral disease in patients with secondary hyperparathyroidism receiving haemodialysis: results of the IMPACT-SHPT study. Nephrol Dial Transplant. 2014 Apr;29(4):899-905. doi: 10.1093/ndt/gfu011. Epub 2014 Feb 4. PMID 24500308
- [Derived] Sharma A, Marshall TS, Khan SS, Johns B. Cost effectiveness of paricalcitol versus cinacalcet with low-dose vitamin D for management of secondary hyperparathyroidism in haemodialysis patients in the USA. Clin Drug Investig. 2014 Feb;34(2):107-15. doi: 10.1007/s40261-013-0151-4. PMID 24214232
- [Derived] Ketteler M, Martin KJ, Wolf M, Amdahl M, Cozzolino M, Goldsmith D, Sharma A, Marx S, Khan S. Paricalcitol versus cinacalcet plus low-dose vitamin D therapy for the treatment of secondary hyperparathyroidism in patients receiving haemodialysis: results of the IMPACT SHPT study. Nephrol Dial Transplant. 2012 Aug;27(8):3270-8. doi: 10.1093/ndt/gfs018. Epub 2012 Mar 2. PMID 22387567

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 272 participants enrolled in the study, 4 did not receive study drug and were not included in the population analyzed.
Groups:
- IV Paricalcitol in the IV Stratum; Cinacalcet in the IV Stratum: IV stratum
- Oral Paricalcitol in the Oral Stratum; Cinacalcet in the Oral Stratum: Oral stratum
Period: Overall Study
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Started | 62 | 64 | 72 | 70
Completed | 50 | 44 | 56 | 53
Not Completed | 12 | 20 | 16 | 17
Not completed — Adverse Event | 2 | 7 | 7 | 7
Not completed — Withdrawal by Subject | 1 | 5 | 1 | 5
Not completed — Protocol Violation | 7 | 3 | 4 | 3
Not completed — Noncompliance | 0 | 2 | 1 | 0
Not completed — Calcium < 7.5 mg/dL on 3 draws | 0 | 0 | 0 | 1
Not completed — Required kidney transplantation | 1 | 3 | 3 | 1
Not completed — Travel for family reasons | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum | Total
Number analyzed (Participants) | 62 | 64 | 72 | 70 | 268
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.71) | 59.9 (12.04) | 65.7 (13.48) | 65.1 (12.50) | 63.1 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 23 | 27 | 100
  Male | 38 | 38 | 49 | 43 | 168
History of type 1 diabetes mellitus [Number; unit: Participants]
  Yes | 6 | 1 | 1 | 2 | 10
  No | 56 | 63 | 71 | 68 | 258
History of type 2 diabetes mellitus [Number; unit: Participants]
  Yes | 37 | 34 | 28 | 9 | 108
  No | 25 | 30 | 44 | 61 | 160
History of angina [Number; unit: Participants]
  Yes | 8 | 2 | 11 | 7 | 28
  No | 54 | 62 | 61 | 63 | 240
History of coronary artery disease [Number; unit: Participants]
  Yes | 25 | 19 | 11 | 6 | 61
  No | 37 | 45 | 61 | 64 | 207
History of left ventricular hypertrophy [Number; unit: Participants]
  Yes | 12 | 4 | 7 | 6 | 29
  No | 50 | 60 | 65 | 64 | 239
History of myocardial infarction [Number; unit: Participants]
  Yes | 12 | 8 | 10 | 8 | 38
  No | 50 | 56 | 62 | 62 | 230

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Achieve a Mean Intact Parathyroid Hormone (iPTH) Value Between 150 to 300 pg/mL During the Evaluation Period (Weeks 21 to 28).
Description: iPTH values obtained during the evaluation period (Weeks 21 to 28) were averaged for each participant with at least 2 iPTH values. Participants whose average iPTH value was between 150 to 300 pg/mL were counted.
Time Frame: Weeks 21 to 28
Population: Randomized participants who received at least 1 dose of study drug and who had both a baseline iPTH value and at least 2 iPTH values during the evaluation period (Weeks 21 to 28)
Measure: Number; unit: Participants
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Number analyzed (Participants) | 52 | 49 | 57 | 53
Participants | 30 | 16 | 31 | 23
Statistical Analysis 1: Comparison: IV Paricalcitol in the IV Stratum vs Cinacalcet in the IV Stratum; With a sample size of 49 participants in each treatment group in the IV stratum, a Fisher's exact test with a 0.050 2-sided significance level will have 81% power to detect a 30% difference in the percentage of participants who achieve iPTH between 150 and 300 pg/mL, assuming the cinacalcet percentage is 36% and the paricalcitol percentage is 66%; Test type: Superiority or Other; p = 0.016, Fisher Exact — No adjustments were made for multiple comparisons between treatment groups since the study was designed to evaluate the primary outcome measure by testing a single hypothesis within each stratum independently
Statistical Analysis 2: Comparison: Oral Paricalcitol in the Oral Stratum vs Cinacalcet in the Oral Stratum; With a sample size of 49 participants in each treatment group in the oral stratum, a Fisher's exact test with a 0.050 2-sided significance level will have 81% power to detect a 30% difference in the percentage of participants who achieve iPTH between 150 and 300 pg/mL, assuming the cinacalcet percentage is 36% and the paricalcitol percentage is 66%; Test type: Superiority or Other; p = 0.260, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants Who Achieve at Least 30% Reduction From Baseline in Intact Parathyroid Hormone (iPTH) as Assessed by the Mean iPTH Obtained During the Evaluation Period (Weeks 21 to 28).
Description: iPTH values obtained during the evaluation period (Weeks 21 to 28) were averaged for each participant with both a baseline iPTH value and at least 2 iPTH values. Participants whose average iPTH value showed a 30% reduction from Baseline were counted.
Time Frame: Weeks 21 to 28
Population: Randomized participants who received at least 1 dose of study drug and who had both a baseline iPTH value at least 2 iPTH values during the evaluation period (Weeks 21 to 28)
Measure: Number; unit: Participants
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Number analyzed (Participants) | 52 | 49 | 57 | 53
Participants | 44 | 24 | 39 | 30
Statistical Analysis 1: Comparison: IV Paricalcitol in the IV Stratum vs Cinacalcet in the IV Stratum; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Oral Paricalcitol in the Oral Stratum vs Cinacalcet in the Oral Stratum; Test type: Superiority or Other; p = 0.239, Fisher Exact

3. Secondary Outcome: Number of Participants Who Achieve at Least 50% Reduction From Baseline in iPTH as Assessed by the Mean iPTH Obtained During the Evaluation Period (Weeks 21 to 28).
Description: iPTH values obtained during the evaluation period (Weeks 21 to 28) were averaged for each participant with both a baseline iPTH value and at least 2 iPTH values. Participants whose average iPTH value showed a 50% reduction from Baseline were counted.
Time Frame: Weeks 21 to 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Number analyzed (Participants) | 52 | 49 | 57 | 53
Participants | 34 | 11 | 26 | 22
Statistical Analysis 1: Comparison: IV Paricalcitol in the IV Stratum vs Cinacalcet in the IV Stratum; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Oral Paricalcitol in the Oral Stratum vs Cinacalcet in the Oral Stratum; Test type: Superiority or Other; p = 0.704, Fisher Exact

4. Secondary Outcome: Analysis of the Number of Participants Who Achieve a Mean iPTH Value Between 150 and 300 pg/mL During the Evaluation Period (Weeks 21 to 28) Using a Cochran-Mantel-Haenszel Test Controlling for IV and Oral Site Randomization Strata
Description: iPTH values obtained during the evaluation period (Weeks 21 to 28) were averaged for each participant with at least 2 iPTH values. Participants whose average iPTH value was between 150 to 300 pg/mL were counted. Data from both the IV and oral strata were analyzed together.
Time Frame: Weeks 21 to 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Number analyzed (Participants) | 52 | 49 | 57 | 53
Participants | 30 | 16 | 31 | 23
Statistical Analysis 1: Comparison: IV Paricalcitol in the IV Stratum vs Cinacalcet in the IV Stratum vs Oral Paricalcitol in the Oral Stratum vs Cinacalcet in the Oral Stratum; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants With Hypocalcemia Defined as < 8.4 mg/dL and Based on the Mean of at Least 2 Values Obtained During the Evaluation Period (Weeks 21 to 28)
Description: Calcium values obtained during the evaluation period (Weeks 21 to 28) were averaged for each participant with at least 2 calcium values. Participants whose average calcium value was < 8.4 mg/dL were counted.
Time Frame: Weeks 21 to 28
Population: Randomized participants who received at least 1 dose of study drug and who had at least 2 calcium values during the evaluation period (Weeks 21 to 28)
Measure: Number; unit: Participants
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Number analyzed (Participants) | 52 | 49 | 56 | 53
Participants | 0 | 23 | 2 | 29
Statistical Analysis 1: Comparison: IV Paricalcitol in the IV Stratum vs Cinacalcet in the IV Stratum; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Oral Paricalcitol in the Oral Stratum vs Cinacalcet in the Oral Stratum; Test type: Superiority or Other; p < 0.001, Fisher Exact

6. Secondary Outcome: Number of Participants With Hypercalcemia Defined as Calcium > 10.5 mg/dL and Based on the Mean of at Least 2 Values Obtained During the Evaluation Period (Weeks 21 to 28)
Description: Calcium values obtained during the evaluation period (Weeks 21 to 28) were averaged for each participant with at least 2 calcium values. Participants whose average calcium value was > 10.5 mg/dL were counted.
Time Frame: Weeks 21 to 28
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Number analyzed (Participants) | 52 | 49 | 56 | 53
Participants | 4 | 0 | 0 | 0
Statistical Analysis 1: Comparison: IV Paricalcitol in the IV Stratum vs Cinacalcet in the IV Stratum; Test type: Superiority or Other; p = 0.118, Fisher Exact
Statistical Analysis 2: Comparison: Oral Paricalcitol in the Oral Stratum vs Cinacalcet in the Oral Stratum; Test type: Superiority or Other; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were reported. These include all adverse events that began on or after the first dose of study drug through 30 days after the last dose of study drug.
Arm/Group | IV Paricalcitol in the IV Stratum | Cinacalcet in the IV Stratum | Oral Paricalcitol in the Oral Stratum | Cinacalcet in the Oral Stratum
Serious Adverse Events (participants affected / at risk) | 22/62 | 28/64 | 22/72 | 15/70
Other Adverse Events (participants affected / at risk) | 48/62 | 46/64 | 59/72 | 54/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Paricalcitol in the IV Stratum (N=62) | Cinacalcet in the IV Stratum (N=64) | Oral Paricalcitol in the Oral Stratum (N=72) | Cinacalcet in the Oral Stratum (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 1 | 0
Atril fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Asthenia (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 1 | 0 | 1
Device occlusion (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 2 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 0 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Brachiocephalic vein stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 1
Vascular stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Venous stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Paricalcitol in the IV Stratum (N=62) | Cinacalcet in the IV Stratum (N=64) | Oral Paricalcitol in the Oral Stratum (N=72) | Cinacalcet in the Oral Stratum (N=70)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 4 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 1 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 4 | 2
Constipation (Gastrointestinal disorders) | 0 | 4 | 2 | 4
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Diarhhoea (Gastrointestinal disorders) | 6 | 5 | 7 | 3
Diverticulum (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 8 | 4 | 7
Vomiting (Gastrointestinal disorders) | 6 | 6 | 9 | 5
Asthenia (General disorders) | 3 | 2 | 1 | 1
Chest pain (General disorders) | 1 | 2 | 3 | 1
Fatigue (General disorders) | 6 | 2 | 1 | 2
Oedema peripheral (General disorders) | 1 | 1 | 2 | 4
Pain (General disorders) | 2 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 4 | 4
Arteriovenous fistula site infection (Infections and infestations) | 2 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 1
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 4 | 2
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4 | 3 | 1 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 2 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 6 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 2 | 0
Blood potassium increased (Investigations) | 0 | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 2 | 2
Haemoglobin decreased (Investigations) | 0 | 3 | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 13 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 8 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 9 | 3 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 1
Dizziness (Nervous system disorders) | 5 | 2 | 1 | 3
Headache (Nervous system disorders) | 3 | 1 | 5 | 2
Hypoaesthesia (Nervous system disorders) | 5 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Hypertension (Vascular disorders) | 6 | 3 | 5 | 4
Hypotension (Vascular disorders) | 8 | 3 | 3 | 1
Steal syndrome (Vascular disorders) | 0 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Using a fixed dosing algorithm based on biochemical criteria may affect interpretation of the results. In the future, the risk/benefit profile of these interventions should be assessed by longer-term clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.